CLINICAL TRIAL: NCT04229056
Title: Computer-Assisted Self-Training to Improve Executive Function Versus Unspecific Training in Patients After Stroke, Cardiac Arrest or in Parkinson's Disease: a Randomized Controlled Trial
Brief Title: COMPuter-assisted Self-training to Improve EXecutive Function
Acronym: COMPEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Glasgow (Other); University of Basel (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Hjernesagen (Unknown); Göteborg University (Other); Aalborg University Hospital (Other); Neurorehabilitering - Kbh, City of Copenhagen (Other)
Responsible Party: Principal Investigator, Hanne Christensen, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19039236
Record Dates: First submitted 2020-01-03; First posted 2020-01-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Stroke; Cardiac Arrest; Cognitive Dysfunction; Executive Dysfunction
Keywords: parkinson disease; stroke; cardiac arrest; executive dysfunction; cognitive dysfunction; computer-based cognitive rehabilitation
MeSH Terms: conditions — Parkinson Disease; Stroke; Heart Arrest; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two parallel groups will be included in this study
Who Masked: Outcomes Assessor
Masking Description: Because of the nature of the intervention, masking participants and investigators is not possible. Outcome assessors will be masked to the group allocation of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specific computer-based cognitive rehabilitation (Experimental): 154 patients will be allocated to specific computer-based cognitive rehabilitation. This group will train with 10 exercises from the cognitive rehabilitation software 'Scientific Brain training PRO'. These 10 exercises are designed to train various executive functions.
  Interventions: Behavioral: Computer-based cognitive rehabilitation (CBCR)
- General computer-based cognitive stimulation (Active Comparator): 154 patients will be allocated to general computer-based cognitive stimulation. This group will train with 10 generally mentally stimulating games on a website specifically designed for this trial. These 10 games are chosen because they are believed to have a low load on executive functions but stimulate over-all concentration and visuoperceptual abilities.
  Interventions: Behavioral: General computer-based cognitive stimulation

INTERVENTIONS:
Behavioral: Computer-based cognitive rehabilitation (CBCR) — CBCR are software-programmes for computers which are clinically developed for rehabilitation of various cognitive functions.
  Arms: Specific computer-based cognitive rehabilitation
Behavioral: General computer-based cognitive stimulation — For this trial we have developed a webpage for general cognitive stimulation, which is designed to provide general computer-based cognitive stimulation.
  Arms: General computer-based cognitive stimulation

SUMMARY:
This project explores the effects of specialized computer-based cognitive rehabilitation (CBCR) targeting executive functions in three groups of patients: Stroke, Cardiac Arrest and Parkinson's Disease. The effect of specialized CBCR is compared to generally cognitively stimulating activities on a computer

DETAILED DESCRIPTION:
This project explores the effects of specialized computer-based cognitive rehabilitation (CBCR) targeting executive functions in three groups of patients: Stroke, Cardiac Arrest and Parkinson's Disease. The effect of specialized CBCR is compared to completing generally cognitively stimulating activities on a computer. A total of 307 patients is expected to be enrolled. All patients will complete a neuropsychological test battery assessing executive functions at inclusion, directly after the eight-week training period and at follow-up three months after the end of the intervention period. Furthermore, all patients will answer questionnaires concerning quality of life and ADL-measures at baseline, after the intervention and at follow-up. All patients will train for a period of 8 weeks, 5 times a week for 60 minutes regardless of their group allocation.

ELIGIBILITY:
Inclusion Criteria:

* A diagnose of stroke, cardiac arrest or Parkinson's disease.
* Aged 18 years or older.
* Impaired working memory measured with CABPad working memory test, cut off for inclusion: 5 symbols or less backwards
* Computer and internet access at home.
* Providing informed consent.

Inclusion criteria specific for stroke

* Inclusion within 6 months post-stroke
* Stroke confirmed by clinical findings and imaging, both AIS and ICH is allowed.
* Initial stroke severity >/= NIHSS 3.

Inclusion criteria specific for cardiac arrest

• Inclusion within 6 months post ictus.

Inclusion criteria specific for Parkinson's disease

* Clinical diagnosis of PD.
* Anti-parkinsonian medical treatment (dopaminergic or other).

Exclusion Criteria:

* Informed consent not provided
* Other neurological or psychiatric disease which is expected to influence the patient's ability to participate in the trial according to the investigator
* Not able to participate according to investigator

Exclusion criteria specific for stroke

* Patients with massive anosognosia for executive dysfunction or patients with no subjective feeling of executive dysfunction (Patient sustains total denial of executive symptoms over time)
* Patients with severe aphasia, in which it is unclear whether the patient's performance on a neuropsychological test-battery is due to aphasia and not executive dysfunction.

Exclusion criteria specific for cardiac arrest • None

Exclusion criteria specific for PD

• Diagnosis of PD Dementia according to the MDS PD Dementia criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
CABPad Working Memory Test | After the end of the intervention (8 weeks after baseline)
  Test of working memory. The higher score the better (theoretically infinite score)

SECONDARY OUTCOMES:
CABPad Working Memory Test - 3 months follow-up | At follow-up visit 3 months after end of intervention
  Test of working memory. The higher score the better (theoretically infinite score)
Minimum Data Set-Home Care- Instrumental Activities of Daily Living (MDS-HC-IADL) | At follow-up visit 3 months after the end of the intervention
  Questionnaire concerning activities of daily living. 0-3 points on an 8-item scale, the fewer points the better.
Trail Making A | Directly after the intervention, eight weeks after inclusion
  Test of processing speed and visual attention. The lower score the better (theoretically infinite score)
Trail Making A | At follow-up visit 3 months after the end of the intervention
  Test of processing speed and visual attention. The lower score the better (theoretically infinite score)
Trail Making B | Directly after the intervention, eight weeks after inclusion
  Test of divided attention, mental flexibility. The lower score the better (theoretically infinite score)
Trail Making B | At follow-up visit 3 months after the end of the intervention
  Test of divided attention, mental flexibility. The lower score the better (theoretically infinite score)
SDMT | Directly after the intervention, eight weeks after inclusion
  Symbol Digit Modalities Test: Test of mental speed. The higher score the better (theoretically infinite score)
SDMT | At follow-up visit 3 months after the end of the intervention
  Symbol Digit Modalities Test: Test of mental speed. The higher score the better (theoretically infinite score)
Phonological verbal fluency test | Directly after the intervention, eight weeks after inclusion
  Test of verbal phonological fluency. The higher score the better (theoretically infinite score)
Phonological verbal fluency test | At follow-up visit 3 months after the end of the intervention
  Test of verbal phonological fluency. The higher score the better (theoretically infinite score)
Categorical verbal fluency test | Directly after the intervention, eight weeks after inclusion
  Test of verbal categorical fluency. The higher score the better (theoretically infinite score)
Categorical verbal fluency test | At follow-up visit 3 months after the end of the intervention
  Test of verbal categorical fluency. The higher score the better (theoretically infinite score)
Fear questionnaire | Directly after the intervention, eight weeks after inclusion
  Questionnaire with 24 items concerning fear on a scale from 0 to 8 where 8 indicates a higher degree of avoidance due to fear
Fear questionnaire | At follow-up visit 3 months after the end of the intervention
  Questionnaire with 24 items concerning fear on a scale from 0 to 8 where 8 indicates a higher degree of avoidance due to fear
mrs: Modified Rankin Scale | Directly after the intervention, eight weeks after inclusion
  Questionnaire concerning disability on a scale from 0 (no symptoms) to 6 (dead): Higher score indicates more severe disability.
mrs: Modified Rankin Scale | At follow-up visit 3 months after the end of the intervention
  Questionnaire concerning disability on a scale from 0 (no symptoms) to 6 (dead). Higher score indicates more severe disability.
IQCODE (Informant Questionnaire on Cognitive Decline in the Elderly) | Directly after the intervention, eight weeks after inclusion
  Cognitive decline in the elderly, reported by partner. A scale of 16 items from 1 (much better) to 5 (much worse). Higher score indicates more severe disability.
IQCODE (Informant Questionnaire on Cognitive Decline in the Elderly) | At follow-up visit 3 months after the end of the intervention
  Cognitive decline in the elderly, reported by partner. A scale of 16 items from 1 (much better) to 5 (much worse). Higher score indicates more severe disability.
EuroQol-5 domain (EQ-5D-5L) | Directly after the intervention, eight weeks after inclusion
  Quality of life scale with 5 domains, each rated from 1-5 indicating slight to severe disability . Higher score indicates more severe disability. Completed by patient and partner
EuroQol-5 domain (EQ-5D-5L) | At follow-up visit 3 months after the end of the intervention
  Quality of life scale with 5 domains, each rated from 1-5 indicating slight to severe disability. Higher score indicates more severe disability. Completed by patient and partner
PDQ 39 (Parkinsons Disease Questionnaire: Only in patients with Parkinson Disease) | Directly after the intervention, eight weeks after inclusion
  Quality of Life questionnaire in patients with Parkinson's Disease. A scale with 39 items rated from 1 (never) to 5 (all the time / Can not do at all). Higher score indicates more severe disability.
PDQ 39 (Parkinsons Disease Questionnaire: Only in patients with Parkinsons Disease) | At follow-up visit 3 months after the end of the intervention
  Quality of Life questionnaire in patients with Parkinson's Disease. A scale with 39 items rated from 1 (never) to 5 (all the time / Can not do at all). Higher score indicates more severe disability.
Compliance | Directly after the intervention, eight weeks after inclusion
  Monitoring of total time spent training in minutes
PHQ-9 (Patient health questionnaire 9) | Directly after the intervention, eight weeks after inclusion
  Questionnaire about health of patient with 9 items rated on a 4 point scale from 0 (not at all) to 3 (almost every day). Higher score indicates more severe disability.
PHQ-9 (Patient health questionnaire 9) | At follow-up visit 3 months after the end of the intervention
  Questionnaire about health of patient with 9 items rated on a 4 point scale from 0 (not at all) to 3 (almost every day). Higher score indicates more severe disability.
2) visual analogue scale (1-10) | Directly after the intervention, eight weeks after inclusion
  After last session: how much they liked doing the training and if they would recommend the intervention to somebody else in their situation. Higher score indicates they liked the training more.
Minimum Data Set-Home Care- Instrumental Activities of Daily Living (MDS-HC-IADL) | Directly after the intervention, eight weeks after inclusion
  Questionnaire concerning activities of daily living. 0-3 points on an 8-item scale, the fewer points the better.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Christensen, Professor, Principal Investigator — Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided
This is currently undecided